CLINICAL TRIAL: NCT05011123
Title: Controlled Study of Immunogenicity and Safety of the Investigational vYF Candidate Vaccine in Comparison to Stamaril in Adults
Brief Title: Study on an Investigational Yellow Fever Vaccine Compared With Stamaril in Adults in Europe and Asia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYF03; U1111-1260-4650 (Registry Identifier: ICTRP); 2022-502047-35 (Registry Identifier: CTIS); 2020-005566-33 (EudraCT Number)
Record Dates: First submitted 2021-08-17; First posted 2021-08-18 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, Sponsor, and Study staff who conduct the safety assessment and the participant will not know which vaccine is administered. Only the study staff who prepare and administer the vaccine and are not involved with the safety evaluation ("vaccinator") will know which vaccine is administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 1 injection of vYF vaccine at Day 1
  Interventions: Biological: Yellow fever vaccine (produced on serum-free Vero cells)
- Group 2 (Active Comparator): 1 injection of Stamaril vaccine at Day 1
  Interventions: Biological: Yellow fever vaccine

INTERVENTIONS:
Biological: Yellow fever vaccine (produced on serum-free Vero cells) — Powder and diluent for suspension for injection - Subcutaneous
  Other Names: vYF vaccine
  Arms: Group 1
Biological: Yellow fever vaccine — Powder and diluent for suspension for injection - Subcutaneous
  Other Names: Stamaril
  Arms: Group 2

SUMMARY:
VYF03 is a phase II, randomized, parallel-group prevention study with 2 arms, active-controlled (Stamaril), observer-blind, multi-center study to assess the non-inferiority of the immune response, in terms of seroconversion rates of the investigational vaccine candidate vYF to the licensed Stamaril, in adults aged 18 years up to 60 years in Europe (EU).

The safety and immunogenicity profile of vYF in a cohort of Asian population of Chinese origin outside of China will also be described. The study will also assess the immunogenicity profiles and the safety profiles of vYF and Stamaril.

Participants will be randomized in a 2:1 ratio to receive a single subcutaneous injection of either the vYF vaccine (380 participants in EU and 80 participants of Chinese origin in Asia) or Stamaril (190 participants in EU and 40 participants of Chinese origin in Asia), on Day 01.

The duration of each participant's participation will be approximately 5 years.

DETAILED DESCRIPTION:
The duration of each participant's participation will be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years up to 60 years* on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile OR Is of childbearing potential and agrees to use an effective contraceptive method (1) or abstinence (1) from at least 4 weeks prior to study intervention administration until at least 4 weeks (2) after study intervention administration.

*18 to 60 years means from the day of the 18th birthday up to the day before the 60th birthday

1. Not applicable for Finland
2. Except for French participants which have to apply 12 weeks contraception after study intervention administration A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) before any dose of study intervention on Day 1 and the test will be repeated on D29 to confirm the participant is still not pregnant within 28 days of vaccine administration.

   - Informed consent form has been signed and dated (3)
3. For participants aged less than 21 years in Singapore, an informed consent form has been signed and dated by both the participant and the parent(s) or another legally acceptable representative

   * Able to attend all scheduled visits and to comply with all study procedures
   * For participants enrolled in Asian countries as part of the additional cohort only: know Chinese origin, defined as having at least one biological parent of Chinese origin, and will be self-reported by the participant

   Exclusion Criteria:

   Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the first 2 years of the 5-year follow-up in another clinical study investigating a vaccine, drug, medical device, or medical procedure. Enrollment in another study after the first 2 years is permitted, assuming that it does not exclude participation in this study.
   * Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination (prior to visit 4), except for influenza vaccination, which may be received at least 2 weeks before study vaccines (4). This exception includes all influenza vaccines including monovalent pandemic influenza vaccines.
   * Previous vaccination against a FV disease at any time including YF with either the study vaccine or another vaccine.
   * Receipt of immune globulins, blood, or blood-derived products in the past 6 months.
   * Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy, or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
   * Known history of any FV infection.
   * Known systemic hypersensitivity to any of the vaccine components, eggs, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
   * Known history or laboratory evidence of HIV infection (5).
   * Known history or laboratory evidence of hepatitis B or hepatitis C infection (6).
   * Personal or family history of thymic pathology (thymoma, thymectomy, or myasthenia).
   * Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
   * Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
   * Chronic illness (7) that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion, including malignancy, such as leukemia, or lymphoma.
   * Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F or 38°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
   * Administration of any anti-viral within 2 months preceding the vaccination and planned administration up to the 6 weeks following the vaccination.
   * Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
   * Planned travel in a YF endemic country within 6 months of investigational or control vaccine administration.
4. Except for Thai participants
5. HIV Serology testing will be performed on all German participants if no evidence of seronegativity in the 90 days preceding vaccination
6. Hepatitis B and Hepatitis C Serology testing will be performed on all German participants if no evidence of seronegativity in the 90 days preceding vaccination
7. Chronic illness may include, but is not limited to, cardiac disorders, renal disorders, auto-immune disorders, diabetes, psychiatric disorders or chronic infection

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 690 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2027-04-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- Finland (3):
  - Investigational Site Number : 2460001, Helsinki
  - Investigational Site Number : 2460002, Tampere
  - Investigational Site Number : 2460003, Turku
- France (6):
  - Investigational Site Number : 2500008, Lyon
  - Investigational Site Number : 2500006, Montpellier
  - Investigational Site Number : 2500001, Nantes
  - Investigational Site Number : 2500007, Nîmes
  - Investigational Site Number : 2500009, Paris
  - Investigational Site Number : 2500004, Pierre-Bénite
- Germany (4):
  - Investigational Site Number : 2760004, Berlin
  - Investigational Site Number : 2760001, Hamburg
  - Investigational Site Number : 2760002, München
  - Investigational Site Number : 2760003, Rostock
- Singapore (3):
  - Investigational Site Number : 7020002, Singapore
  - Investigational Site Number : 7020003, Singapore
  - Investigational Site Number : 7020001, Singapore
- Spain (4):
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Barcelona
- Thailand (3):
  - Investigational Site Number : 7640001, Bangkok
  - Investigational Site Number : 7640002, Bangkok
  - Investigational Site Number : 7640003, Nonthaburi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 23 sites in 6 countries in Europe and Asia from 07 October 2021 to 25 April 2022. Interim results are presented up to Year 2 follow-up, data base lock (DBL) date of 01 August 2024.
Pre-assignment Details: A total of 690 participants were randomized in a 2:1 ratio to receive a single subcutaneous (SC) injection of either yellow fever vaccine (vYF) vaccine or Stamaril. A subset of participants enrolled in European Union (EU) and Asia at selected sites provided an additional post-vaccination blood sample on Day 11 to assess the early immune response elicited by both vaccines in terms of neutralizing antibody (Nab) titers.
Groups:
- vYF 0.5 mL: Participants received 1 dose of vYF vaccine 0.5 milliliter (mL) as a SC injection on Day 1.
- Stamaril 0.5 mL: Participants received 1 dose of Stamaril vaccine 0.5 mL as a SC injection on Day 1.
Period: Overall Study
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Started | 455 | 235
Randomized and Vaccinated | 454 | 235
Completed | 407 | 217
Not Completed | 48 | 18
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 7 | 6
Not completed — Ongoing at the time of DBL date | 36 | 10
Not completed — Randomized but did not receive vaccination | 1 | 0

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants with data in the case report form (CRF).
Groups:
- vYF 0.5 mL: Participants received 1 dose of vYF vaccine 0.5 mL as a SC injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL | Total
Number analyzed (Participants) | 455 | 235 | 690
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (11.76) | 37.1 (11.51) | 37.1 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 136 | 389
  Male | 202 | 99 | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 85 | 43 | 128
  Black or African American | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 356 | 187 | 543
  Multiple origin | 3 | 2 | 5
  Not Reported | 2 | 0 | 2
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Yellow Fever-naive Participants Who Achieved Seroconversion 28 Days Post Dose 1 Enrolled in European Union
Description: Seroconversion was defined as a 4-fold increase in Nab titers as compared to the pre-vaccination value. YF-naive participants (or negative) at baseline corresponded to participants with no detectable YF Ab titers before vaccination. The YF NAb titers were determined using a validated live virus microneutralization (MN) assay. Percentages are rounded off to the tenth decimal place.
Time Frame: 28 days post dose 1 (Day 29)
Population: The per-protocol analysis set (PPAS) was a subset of the full analysis set (FAS). The FAS included the subset of randomized participants who received at least 1 dose of the study vaccine or control vaccine and had a valid post-vaccination blood sample result. Only YF-naive participants enrolled in EU with data collected are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 322 | 160
percentage of participants | 98.1 [96.0 to 99.3] | 99.4 [96.6 to 100]
Statistical Analysis 1: Comparison: vYF 0.5 mL vs Stamaril 0.5 mL; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) was >-5%; Difference in percentage of participants = -1.2, 95% CI 2-sided [-3.4 to 1.8] — 95% CI of the difference was calculated from the Wilson score method without continuity correction

2. Secondary Outcome: Percentage of Participants Who Achieved Seroconversion 28 Days Post Dose 1 Enrolled in European Union
Description: Seroconversion was defined as a 4-fold increase in Nab titers as compared to the pre-vaccination value. The YF NAb titers were determined using a validated live virus MN assay. Percentages are rounded off to the tenth decimal place.
Time Frame: 28 days post dose 1 (Day 29)
Population: The FAS included the subset of randomized participants who received at least 1 dose of the study vaccine or control vaccine and had a valid post-vaccination blood sample result. Only participants enrolled in EU with data collected are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 369 | 190
percentage of participants | 95.9 [93.4 to 97.7] | 96.8 [93.3 to 98.8]
Statistical Analysis 1: Comparison: vYF 0.5 mL vs Stamaril 0.5 mL; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-5%; Difference in percentage of participants = -0.9, 95% CI 2-sided [-4.0 to 3.0] — 95% CI of the difference was calculated from the Wilson score method without continuity correction

3. Secondary Outcome: Percentage of Participants Who Achieved Seroconversion Enrolled in European Union and Asia
Description: Seroconversion was defined as a 4-fold increase in Nab titers as compared to the pre-vaccination value: as compared to the Day 1 titers at each timepoint up to Month 6; as compared to the last planned previous timepoint from Year 1 onwards. The YF NAb titers were determined using a validated live virus MN assay. Percentages are rounded off to the tenth decimal place.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: FAS: subset of randomized participants who received at least 1 dose of study vaccine or control vaccine and had a valid post-vaccination blood sample result. Day 11: subset of participants enrolled in EU and Asia at selected sites who provided an additional post-vaccination blood sample on Day 11 to assess early immune response elicited by both vaccines in terms of Nab titers. Only participants enrolled in EU and Asia with data collected at specified timepoints are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 369 | 190
percentage of participants
  EU: Day 11: number analyzed (Participants) | 56 | 33
  EU: Day 11 | 30.4 [18.8 to 44.1] | 63.6 [45.1 to 79.6]
  EU: Day 29 | 95.9 [93.4 to 97.7] | 96.8 [93.3 to 98.8]
  EU: Month 6: number analyzed (Participants) | 360 | 187
  EU: Month 6 | 95.8 [93.2 to 97.6] | 95.2 [91.1 to 97.8]
  EU: Year 1: number analyzed (Participants) | 340 | 183
  EU: Year 1 | 3.2 [1.6 to 5.7] | 4.4 [1.9 to 8.4]
  EU: Year 2: number analyzed (Participants) | 321 | 169
  EU: Year 2 | 0.9 [0.2 to 2.7] | 3.0 [1.0 to 6.8]
  Asia: Day 11: number analyzed (Participants) | 39 | 21
  Asia: Day 11 | 5.1 [0.6 to 17.3] | 33.3 [14.6 to 57.0]
  Asia: Day 29: number analyzed (Participants) | 78 | 42
  Asia: Day 29 | 87.2 [77.7 to 93.7] | 97.6 [87.4 to 99.9]
  Asia: Month 6: number analyzed (Participants) | 77 | 39
  Asia: Month 6 | 85.7 [75.9 to 92.6] | 100 [91.0 to 100]
  Asia: Year 1: number analyzed (Participants) | 76 | 38
  Asia: Year 1 | 1.3 [0 to 7.1] | 0 [0 to 9.3]
  Asia: Year 2: number analyzed (Participants) | 75 | 40
  Asia: Year 2 | 1.3 [0 to 7.2] | 2.5 [0.1 to 13.2]

4. Secondary Outcome: Percentage of Participants Who Achieved Seroprotection to Yellow Fever Virus Enrolled in European Union and Asia
Description: Seroprotection was defined as NAb titers >=threshold of 10 (1/dilution). YF-naive participants (or negative) at baseline corresponded to participants with no detectable YF Ab titers before vaccination. The YF NAb titers were determined using a validated live virus MN assay. Percentages are rounded off to the tenth decimal place.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 371 | 190
percentage of participants
  EU: Day 1 | 4.3 [2.5 to 6.9] | 7.9 [4.5 to 12.7]
  EU: Day 11: number analyzed (Participants) | 56 | 33
  EU: Day 11 | 48.2 [34.7 to 62.0] | 81.8 [64.5 to 93.0]
  EU: Day 29: number analyzed (Participants) | 369 | 190
  EU: Day 29 | 98.6 [96.9 to 99.6] | 99.5 [97.1 to 100]
  EU: Month 6: number analyzed (Participants) | 360 | 187
  EU: Month 6 | 98.1 [96.0 to 99.2] | 100 [98.0 to 100]
  EU: Year 1: number analyzed (Participants) | 341 | 185
  EU: Year 1 | 98.5 [96.6 to 99.5] | 99.5 [97.0 to 100]
  EU: Year 2: number analyzed (Participants) | 327 | 170
  EU: Year 2 | 98.5 [96.5 to 99.5] | 100 [97.9 to 100]
  Asia: Day 1: number analyzed (Participants) | 78 | 42
  Asia: Day 1 | 6.4 [2.1 to 14.3] | 7.1 [1.5 to 19.5]
  Asia: Day 11: number analyzed (Participants) | 39 | 21
  Asia: Day 11 | 28.2 [15.0 to 44.9] | 66.7 [43.0 to 85.4]
  Asia: Day 29: number analyzed (Participants) | 78 | 42
  Asia: Day 29 | 96.2 [89.2 to 99.2] | 100 [91.6 to 100]
  Asia: Month 6: number analyzed (Participants) | 77 | 39
  Asia: Month 6 | 96.1 [89.0 to 99.2] | 100 [91.0 to 100]
  Asia: Year 1: number analyzed (Participants) | 77 | 40
  Asia: Year 1 | 94.8 [87.2 to 98.6] | 100 [91.2 to 100]
  Asia: Year 2: number analyzed (Participants) | 75 | 40
  Asia: Year 2 | 96.0 [88.8 to 99.2] | 100 [91.2 to 100]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Yellow Fever Virus in Participants Enrolled in European Union and Asia
Description: GMTs of antibody against YF virus was measured using a validated live virus MN assay.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 371 | 190
titer
  EU: Day 1 | 5.62 [5.29 to 5.98] | 6.18 [5.52 to 6.92]
  EU: Day 11: number analyzed (Participants) | 56 | 33
  EU: Day 11 | 26.6 [14.4 to 49.2] | 52.3 [29.8 to 91.5]
  EU: Day 29: number analyzed (Participants) | 369 | 190
  EU: Day 29 | 2229 [1928 to 2577] | 1060 [884 to 1270]
  EU: Month 6: number analyzed (Participants) | 360 | 187
  EU: Month 6 | 562 [493 to 641] | 425 [365 to 495]
  EU: Year 1: number analyzed (Participants) | 341 | 185
  EU: Year 1 | 454 [391 to 527] | 420 [353 to 499]
  EU: Year 2: number analyzed (Participants) | 327 | 170
  EU: Year 2 | 310 [268 to 359] | 349 [292 to 416]
  Asia: Day 1: number analyzed (Participants) | 78 | 42
  Asia: Day 1 | 6.16 [5.13 to 7.39] | 5.63 [4.83 to 6.57]
  Asia: Day 11: number analyzed (Participants) | 39 | 21
  Asia: Day 11 | 10.3 [6.36 to 16.7] | 16.6 [10.0 to 27.7]
  Asia: Day 29: number analyzed (Participants) | 78 | 42
  Asia: Day 29 | 1204 [792 to 1831] | 1167 [843 to 1616]
  Asia: Month 6: number analyzed (Participants) | 77 | 39
  Asia: Month 6 | 495 [355 to 690] | 398 [300 to 527]
  Asia: Year 1: number analyzed (Participants) | 77 | 40
  Asia: Year 1 | 303 [209 to 438] | 245 [174 to 344]
  Asia: Year 2: number analyzed (Participants) | 75 | 40
  Asia: Year 2 | 168 [127 to 223] | 143 [104 to 196]

6. Secondary Outcome: Geometric Mean Titers Ratio (GMTRs) of Antibodies Against Yellow Fever Virus in Participants Enrolled in European Union and Asia
Description: GMTs of antibody against YF virus was measured using a validated live virus MN assay. Ratio was calculated as post-vaccination titer at Days 11, 29 and Month 6 to pre-vaccination titer at Day 1; post-vaccination titer at Year 1 to pre-vaccination titer at Month 6; post-vaccination titer at Year 2 to pre-vaccination titer at Year 1.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 369 | 190
ratio
  EU: Day 11/Day 1: number analyzed (Participants) | 56 | 33
  EU: Day 11/Day 1 | 3.12 [1.85 to 5.27] | 4.92 [3.02 to 8.03]
  EU: Day 29/Day 1 | 206 [176 to 241] | 90.9 [74.1 to 111]
  EU: Month 6/Day 1: number analyzed (Participants) | 360 | 187
  EU: Month 6/Day 1 | 52.3 [45.5 to 60.0] | 36.7 [30.7 to 43.9]
  EU: Year 1/Month 6: number analyzed (Participants) | 340 | 183
  EU: Year 1/Month 6 | 0.810 [0.738 to 0.889] | 0.993 [0.884 to 1.11]
  EU: Year 2/Year 1: number analyzed (Participants) | 321 | 169
  EU: Year 2/Year 1 | 0.655 [0.597 to 0.718] | 0.822 [0.716 to 0.944]
  Asia: Day 11/Day 1: number analyzed (Participants) | 39 | 21
  Asia: Day 11/Day 1 | 1.31 [1.04 to 1.65] | 2.05 [1.36 to 3.08]
  Asia: Day 29/Day 1: number analyzed (Participants) | 78 | 42
  Asia: Day 29/Day 1 | 105 [67.0 to 164] | 109 [75.9 to 156]
  Asia: Month 6/Day 1: number analyzed (Participants) | 77 | 39
  Asia: Month 6/Day 1 | 43.1 [30.0 to 61.7] | 36.9 [27.4 to 49.8]
  Asia: Year 1/Month 6: number analyzed (Participants) | 76 | 38
  Asia: Year 1/Month 6 | 0.607 [0.497 to 0.741] | 0.601 [0.474 to 0.762]
  Asia: Year 2/Year 1: number analyzed (Participants) | 75 | 40
  Asia: Year 2/Year 1 | 0.542 [0.452 to 0.649] | 0.585 [0.470 to 0.729]

7. Secondary Outcome: Number of Participants With Unsolicited Systemic Adverse Events (AEs)
Description: An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, ie, pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to 30 minutes post vaccination on Day 1
Population: The safety analysis set (SafAS) included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 454 | 235
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. An injection site reaction was an AR at and around the injection site of the study vaccine.
Time Frame: Up to 7 days post vaccination (Day 8)
Population: The SafAS included all participants who received at least 1 dose of the study vaccines. Only participants with data collected are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 450 | 233
Participants | 152 | 50

9. Secondary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. Solicited systemic reactions were systemic AEs observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF.
Time Frame: Up to 14 days post vaccination (Day 15)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 450 | 233
Participants | 222 | 126

10. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: as for outcome 7
Time Frame: Up to 28 days post vaccination (Day 29)
Population: The SafAS included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 454 | 235
Participants | 138 | 68

11. Secondary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) up to 6 Months Post-Vaccination
Description: An SAE was any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor could be appropriate. AESIs included serious hypersensitivity/allergic reactions, organ failure/serious viscerotropic events, serious neurologic events.
Time Frame: From the first dose of study vaccine administration (Day 1) up to 6 months post vaccination, approximately up to Day 181
Population: The SafAS included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 454 | 235
Participants
  SAEs | 6 | 8
  AESIs | 0 | 1

12. Secondary Outcome: Number of Participants With Serious Adverse Events and Deaths up to Day 1030
Description: An SAE was any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: From the first dose of study vaccine administration (Day 1) up to DBL date of 01 August 2024, approximately up to Day 1030
Population: The SafAS included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
Number analyzed (Participants) | 454 | 235
Participants
  SAEs | 11 | 11
  Deaths | 0 | 0

13. Secondary Outcome: Number of Participants With Serious Adverse Events and Deaths Up to Year 5
Description: as for outcome 12
Time Frame: From the first dose of study vaccine administration (Day 1) up to end of study, approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-04

ADVERSE EVENTS:
Time Frame: AEs, SAEs and all-cause mortality (deaths) were collected from the first dose of study vaccine administration (Day 1) up to DBL date of 01 August 2024, approximately up to Day 1030.
Description: Analysis was performed on the SafAS. Interim results are presented up to Year 2 follow-up, DBL date of 01 August 2024.
Arm/Group | vYF 0.5 mL | Stamaril 0.5 mL
All-Cause Mortality (participants affected / at risk) | 0/454 | 0/235
Serious Adverse Events (participants affected / at risk) | 11/454 | 11/235
Other Adverse Events (participants affected / at risk) | 266/454 | 141/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vYF 0.5 mL (N=454) | Stamaril 0.5 mL (N=235)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 3 (3)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Benign Neoplasm Of Testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vYF 0.5 mL (N=454) | Stamaril 0.5 mL (N=235)
Injection Site Erythema (General disorders) | 30 (30) | 1 (1)
Injection Site Pain (General disorders) | 144 (144) | 49 (49)
Malaise (General disorders) | 105 (105) | 61 (61)
Myalgia (Musculoskeletal and connective tissue disorders) | 123 (123) | 65 (65)
Headache (Nervous system disorders) | 168 (168) | 99 (99)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT05011123/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT05011123/SAP_001.pdf